CLINICAL TRIAL: NCT00001171
Title: Evaluation of Biological, Immunological and Therapeutic Parameters in Brain Tumor Patients
Brief Title: Evaluation of Factors in Human Brain Tumors
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 790089; 79-N-0089
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-09

CONDITIONS: Brain Neoplasm; Glioblastoma; Glioma; Pituitary Neoplasm
Keywords: Brain Tumors; Glioma; Glioblastoma Multiforme; Pituitary Adenoma
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Glioma; Pituitary Neoplasms

SUMMARY:
Presently, patients with primary malignant brain tumors have a life expectancy of 15 weeks following surgery unless they receive additional types of therapy (chemotherapy, radiotherapy, and/or immunotherapy). Patients that receive additional therapy can increase life expectancy to 50 weeks.

The statistics on the life expectancy and survival have increased efforts among researchers to develop new treatments for primary malignant brain tumors.

This research project involves the growth and study of human brain tumor cells outside the body in the laboratory as part of an attempt to better understand these tumors and to develop more effective treatments for them.

DETAILED DESCRIPTION:
This protocol involves the study of human brain tumor cells outside the body in the laboratory as part of an attempt to better understand these tumors and to develop more effective therapeutic measures.

Malignant primary brain tumor patients at present have a life expectancy of approximately 15 weeks following surgery unless other adjunctive measures are taken. With currently available adjunctive therapy the life expectancy reaches 50 weeks.

These survival data have spurred extensive efforts to develop new treatment modalities. Radiation, chemotherapy and immunotherapy have been mildly helpful adjuncts but their use has been largely on empirical grounds or on the basis of experimentation on animal tumor models often quite different in nature from human brain tumors.

Our group has sought to develop data upon which to devise new treatment strategies for patients with malignant brain tumors.

The foundation of our approach rests upon the use of in vitro studies of the cell biology of each patient's tumor.

It is our plan to utilize these tumors for in vitro investigation of the immunology, biology, biochemistry and molecular biology of brain tumors. Optimal conventional therapy will be given to the patients as we seek to learn more of how the scientific information obtained can be used to help them.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients to be studied will have either undergone surgical confirmation of a malignant primary brain tumor or be considered likely to have that diagnosis on the basis of diagnostic studies.

They should have survival likelihood of at least three months and be able to comprehend the nature of the proposed program.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800
Dates: Start 1979-07; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Manski TJ, Heffner DK, Glenn GM, Patronas NJ, Pikus AT, Katz D, Lebovics R, Sledjeski K, Choyke PL, Zbar B, Linehan WM, Oldfield EH. Endolymphatic sac tumors. A source of morbid hearing loss in von Hippel-Lindau disease. JAMA. 1997 May 14;277(18):1461-6. doi: 10.1001/jama.277.18.1461. PMID 9145719
- [Background] Mason RB, Nieman LK, Doppman JL, Oldfield EH. Selective excision of adenomas originating in or extending into the pituitary stalk with preservation of pituitary function. J Neurosurg. 1997 Sep;87(3):343-51. doi: 10.3171/jns.1997.87.3.0343. PMID 9285597
- [Background] Zunkeler B, Carson RE, Olson J, Blasberg RG, Girton M, Bacher J, Herscovitch P, Oldfield EH. Hyperosmolar blood-brain barrier disruption in baboons: an in vivo study using positron emission tomography and rubidium-82. J Neurosurg. 1996 Mar;84(3):494-502. doi: 10.3171/jns.1996.84.3.0494. PMID 8609564